CLINICAL TRIAL: NCT01206049
Title: Randomized Phase II Trial of Combination Chemotherapy With Panitumumab or Bevacizumab for Patients With Inoperable Cholangiocarcinoma Without KRAS Mutations
Brief Title: Combination Chemotherapy Plus Panitumumab or Bevacizumab for Inoperable Cholangiocarcinoma Without KRAS Mutations
Acronym: GOC-B-P
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010-020385-13
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2016-06

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Inoperable; KRAS mutation; Biological treatment; Combination chemotherapy; Monoclonal antibody
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine; Oxaliplatin; Capecitabine; Panitumumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination chemotherapy + panitumumab (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Panitumumab
- Combination chemotherapy + bevacizumab (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine — 1,000 mg/m2 on day 1 of a 2 weeks cycle
Drug: Oxaliplatin — 60 mg/m2 on day 1 of a 2 weeks cycle
Drug: Capecitabine — 1,000 mg/m2 x 2 daily on days 1-7 of a 2 weeks cycle
Drug: Panitumumab — 6 mg/kg on day 1 of a 2 weeks cycle
  Arms: Combination chemotherapy + panitumumab
Drug: Bevacizumab — 10 mg/kg on day 1 of a 2 weeks cycle
  Arms: Combination chemotherapy + bevacizumab

SUMMARY:
The purpose of this study is to determine the rate of progression free survival of patients with inoperable cholangiocarcinoma 6 months after enrollment in the study. The patients are treated with combination chemotherapy supplemented by biological agents panitumumab or bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma arisen from gall bladder, extra- or intrahepatic bile ducts or malignant cells consistent with the above and simultaneous radiologic findings consistent with cholangiocarcinoma
* Minimum 18 years of age
* Curative treatment currently not an option (operation, stereotactic radiation treatment or similar)
* KRAS analyzed and found wild-type (wt)
* Performance status 0-2
* Evaluable disease according to RECIST, i.e. the disease need not be measurable
* Hematology: ANC ≥1.5x10^9/l. Thrombocytes ≥ 100x10^9/l
* Biochemistry: Bilirubinemia ≤ 3 x upper normal level. ALAT ≤ 5 x upper normal level.
* Creatinine ≤ upper normal level. At raised creatinine level the measured or calculated GFR must be at least 50% of the lower normal level
* Fertile women must present a negative pregnancy test and use secure birth control during and 6 months after treatment. Men with fertile partners must also take care of secure birth control.
* Written and orally informed consent

Exclusion Criteria:

* Previous cytostatic treatment of inoperable cholangiocarcinoma
* Adjuvant or neoadjuvant chemotherapy, radiation therapy or immunotherapy within 4 weeks prior to treatment start
* Other concomitant experimental treatment
* Severe medical disease such as considerable heart disease, serious active infection or other disease making the patient unfit for study participation as assessed by investigator
* Other malignant disease within 5 years prior to enrolment except from non-melanotic skin cancer and carcinoma in situ cervicis uteri
* Interstitial pneumonitis or subsequent pulmonary fibrosis
* Pregnant or breastfeeding women
* Large-scale surgical intervention, excision biopsy or significant traumatic lesions within 28 days prior to treatment start or presumption that large-scale surgery will become necessary during study treatment.
* Significant non-healing wound or ulcers
* Active hemorrhage or increased risk of hemorrhage (e.g. tumor invasion in large vessels or known esophagus varices)
* Known hypersensitivity to panitumumab, bevacizumab or any of the auxiliary agents
* Grade IV fistulas
* Uncontrolled hypertension, i.e. symptomatic hypertension or non-medically stabilized hypertension >160/100
* Haemoptysis > 2.5 ml within 2 weeks prior to enrolment
* Previous serious and unexpected reactions or know hypersensitivity to two or more of the applied cytostatics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The fraction of patients alive and without progression at 6 months | 6 months from enrollment date

SECONDARY OUTCOMES:
Response rate before cross-over | 6 months after enrollment or earlier in case of progression
Overall survival | 6 months
Progression free survival and response rate after cross-over | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, MD, DMSc, Study Chair — Department of Oncology, Vejle Hospital
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark